CLINICAL TRIAL: NCT04317963
Title: Real-world Evaluation of Bezlotoxumab for the Management of Clostridioides Difficile Infection
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Eric R Wenzler, Assistant Professor, Department of Pharmacy Practice, University of Illinois at Chicago
Other Study IDs: 2019-1381
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Clostridium Difficile Infection; Clostridium Difficile Infection Recurrence
MeSH Terms: conditions — Clostridium Infections | interventions — bezlotoxumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Cases: Patients who have received bezlotoxumab 10 mg/kg intravenously in addition to standard CDI treatment.
  Interventions: Biological: Bezlotoxumab
- Controls: Patients who have received only standard CDI treatment.
  Interventions: Drug: Standard CDI treatment

INTERVENTIONS:
Biological: Bezlotoxumab — Bezlotoxumab 10 mg/kg IV infusion in addition to standard CDI treatment
  Groups: Cases
Drug: Standard CDI treatment — Standard CDI treatment includes one or a combination of oral vancomycin, oral vancomycin taper and/or pulse, fidaxomicin, and fidaxomicin taper and/or pulse
  Groups: Controls

SUMMARY:
This is a retrospective case:control study examining the use of adjunctive bezlotoxumab to standard C. difficile infection (CDI) treatment compared to standard CDI treatment alone in patients with CDI seen in an academic medical center's specialty outpatient clinic.

DETAILED DESCRIPTION:
This specialty clinic is a unique practice setting where patients with ≥1 recurrent CDI and/or refractory disease are referred. The study will represent real-world data on the clinical use of bezlotoxumab as adjunctive therapy in combination with vancomycin or fidaxomicin for the treatment of patients with recurrent CDI. Retrospective chart review will be conducted for patients who visited the specialty CDI clinic between 1/1/2005 through 12/5/2019. Case patients will be defined as patients who have received bezlotoxumab 10 mg/kg intravenously in addition to standard CDI treatment. Controls will be defined as patients who have received only standard CDI treatment and will be enrolled in a 2:1 ratio to cases. The primary outcome is recurrence of CDI. Recurrence is defined as a new episode of C. difficile infection that occurs after the initial clinical cure of the baseline episode within 12 weeks of receipt of bezlotoxumab or standard CDI treatment. Clinical cure is defined as no diarrhea for 2 consecutive days after completion of standard-of-care CDI therapy. Recurrent CDI will be diagnosed via clinical signs and symptoms and CDI diagnostic assay.

ELIGIBILITY:
Inclusion Criteria (Cases):

* Age 18 years and older
* Diagnosis of C. difficile infection by clinical signs and symptoms and/or C. difficile diagnostic assay
* Received bezlotoxumab in addition to standard CDI treatment

Inclusion Criteria (Controls):

* Age 18 years and older
* Diagnosis of C. difficile infection by clinical signs and symptoms and/or C. difficile diagnostic assay
* Received only standard CDI treatment

Exclusion Criteria:

* Diarrhea due to causes other than C. difficile
* Incomplete documentation in the electronic medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated for C. difficile infection
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Rate of CDI Recurrence | within 12 weeks of receipt of bezlotoxumab
  New episode of C. difficile infection that occurs after initial clinical cure of the baseline episode within 12 weeks of receipt of bezlotoxumab or completion of standard CDI treatment.

SECONDARY OUTCOMES:
Clinical cure | 2 consecutive days after completion of standard-of-care CDI therapy.
  Clinical cure is defined as no diarrhea for 2 consecutive days after completion of standard-of-care CDI therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Wenzler, PharmD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States